CLINICAL TRIAL: NCT07000006
Title: The Effect of Exercise on Low Back Pain and Quality of Life in Peritoneal Dialysis Patients: a Randomized Controlled Trial
Brief Title: The Effect of Exercise on Low Back Pain in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA25PD-2-02
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: End Stage Renal Disease (ESRD); Peritoneal Dialysis Complication
Keywords: Home-based Exercise; Core Stability; Low Back Pain; Peritoneal Dialysis; Physical Function
MeSH Terms: conditions — Kidney Failure, Chronic; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional test. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants in the intervention group will receive a personalized home-based exercise program focused on core muscle strength and trunk stability during dialysis days. Each session will last 40 to 45 minutes, 3 times per week, over 12 weeks (36 sessions total). Sessions will be conducted synchronously via a teleconference application (e.g., Google Meet), with professionals supervising and controlling participant access.
  Interventions: Behavioral: Home-based Core Stability Exercise
- Control group (No Intervention): Patients in the control group will continue receiving standard nephrological care. Over the 12-week study period, they will be instructed to maintain their usual treatment routines, physical activity, and diet patterns.

INTERVENTIONS:
Behavioral: Home-based Core Stability Exercise — The online exercise program aims to improve trunk stability and reduce low back pain. A clinical exercise physiologist will deliver real-time exercise sessions, with each session lasting 40-45 minutes, three days a week for 12 weeks. Participants will join private group sessions using a free video platform.
  Arms: Exercise group

SUMMARY:
The goal of this randomized controlled trial is to find out if exercise can help reduce low back pain and improve quality of life in people receiving peritoneal dialysis (PD). The main questions it aims to answer are:

Does a structured exercise program lower low back pain in PD participants?

Does exercise improve their health-related quality of life?

Researchers will compare a group of participants who do regular exercises with a group who receive usual care, to see if the exercises make a difference.

Participants will:

Join a home-based exercise program designed for people on PD.

Follow the program for a specific period while continuing their dialysis treatment.

Complete assessments on their pain and quality of life before and after the intervention.

DETAILED DESCRIPTION:
The effect of exercise on low back pain and quality of life in peritoneal dialysis patients: a randomized controlled trial Pain represents a significant burden for patients undergoing peritoneal dialysis (PD), with recent research indicating an incidence rate of approximately 33.1% in this population. This prevalence notably exceeds the 20% reported in the general adult population. While PD offers several advantages over hemodialysis-including greater autonomy and improved initial quality of life-patients often face significant musculoskeletal complications, particularly low back pain (LBP). LBP in PD patients is multifactorial, arising from altered body mechanics due to dialysate instillation, pre-existing spinal pathology, sedentary lifestyle, and muscular weakness. Recent studies indicate that over 60% of patients on chronic PD experience LBP, which may be exacerbated by factors such as advanced age, increased body mass index, and comorbidities. This pain is not only a source of physical discomfort but also contributes to reduced mobility, increased disability, and a marked decline in health-related quality of life (HRQOL).

The etiology of low back pain in PD patients appears multifactorial, potentially stemming from altered biomechanics related to the peritoneal dialysis process, disruptions in bone mineral metabolism, and physiological changes associated with kidney disease. Research has demonstrated that pain in this population is independently associated with depressive symptoms, poor sleep quality, and reduced quality of life. The continuous presence of dialysate fluid in the peritoneal cavity may alter spinal alignment and stress load distribution, potentially contributing to musculoskeletal discomfort and pain.

The potential causes of pain in PD patients include disruption in bone mineral density, muscular deconditioning, and mechanical stressors related to the dialysis procedure itself. The presence of dialysate in the peritoneal cavity can alter abdominal mechanics and potentially contribute to low back pain through changes in posture and movement patterns. Furthermore, PD patients are generally physically inactive and frail, which may exacerbate existing musculoskeletal conditions.

Case reports have documented severe manifestations of spinal issues in PD patients, including spondylodiscitis presenting with arm and neck pain. While these represent extreme cases, they highlight the vulnerability of the musculoskeletal system in this patient population. Female PD patients particularly report higher pain severity and interference levels, suggesting gender-specific considerations may be necessary when addressing pain management strategies.

Pain severity in PD patients has been found to negatively correlate with supplement doses for vitamin D3 and calcium, indicating complex interactions between pain perception, bone health, and mineral metabolism. These relationships suggest that interventions targeting musculoskeletal health, such as structured exercise programs, may potentially address multiple factors contributing to pain in this population.

Quality of life is a critical outcome in the management of PD patients, as it encompasses physical, psychological, and social well-being. Evidence consistently shows that pain, particularly LBP, is closely linked to lower HRQOL scores, affecting patients' ability to perform daily activities, maintain employment, and engage socially. Although PD is generally associated with better HRQOL compared to hemodialysis, the burden of chronic pain and physical limitations remains substantial, often leading to increased healthcare utilization and diminished patient autonomy. Interventions that can alleviate pain and enhance physical function are thus of paramount importance for this population.

Despite the recognized prevalence and impact of LBP in PD patients, there is a notable gap in the literature regarding effective, accessible interventions tailored to their unique needs. While exercise programs have demonstrated benefits in reducing pain and improving function in the general population and in patients with CKD, few studies have rigorously evaluated home-based exercise interventions specifically targeting core muscle strength and trunk stability in PD patients. Moreover, the feasibility and efficacy of such programs in improving both pain outcomes and overall quality of life have not been adequately explored, especially in the context of randomized controlled trials.

This study aims to address these gaps by evaluating the effect of a structured, home-based exercise intervention focusing on core muscle strength and trunk stability on LBP and quality of life in peritoneal dialysis patients.

The rationale for this study is grounded in the urgent need for evidence-based, scalable interventions that can be implemented in the home setting to improve pain and quality of life in PD patients. The investigators hypothesize that a home-based exercise program focusing on core stability will significantly reduce pain severity and enhance HRQOL compared to standard care, with additional benefits in physical function and symptom burden. By rigorously evaluating this intervention in a randomized controlled trial, this study seeks to provide critical evidence to inform clinical practice and improve outcomes for this vulnerable population.

The investigators hypothesize that:

1. PD patients who participate in the 12-week home-based exercise program will experience greater reductions in low back pain, as measured by the Brief Pain Inventory (BPI), compared to the control group receiving standard care.
2. PD patients in the intervention group will demonstrate greater improvements in quality of life, as measured by the SF-36 questionnaire, compared to the control group.
3. The exercise program will lead to improvements in physical function and associated secondary outcomes, and will be feasible and safe for implementation among PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* On peritoneal dialysis for at least 6 months
* Reported chronic low back pain for ≥3 months
* Medically stable with physician approval for exercise
* Ability to provide informed consent
* Access to a smart device and internet connection
* Cognitive ability to follow instructions and participate in virtual sessions

Exclusion Criteria:

* Unstable cardiovascular conditions (e.g., recent MI, angina)
* Active infections or acute illness
* Severe musculoskeletal limitations or recent orthopedic surgery
* Neurological disorders impairing mobility
* Severe dyspnea at rest or during ADLs (NYHA Class IV)
* Participation in regular exercise programs ≥3 times/week targeting core strength
* Psychiatric or cognitive impairment interfering with participation
* Recent hospitalization for back surgery or spine-related intervention within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain Severity | Baseline, Week 6 (mid-intervention), and Week 12 (post-intervention)]
  Pain severity will be assessed using the Brief Pain Inventory (BPI), which includes four 0-10 numeric rating scales measuring worst, least, average, and current pain over the past 24 hours. Higher scores indicate greater pain severity. A reduction of at least 2 points on the average pain scale is considered clinically meaningful. Assessments will follow standardized BPI administration protocols validated in renal and chronic pain populations.
Change in Health-Related Quality of Life | Baseline and Week 12
  Quality of life will be measured using the Short Form-36 Health Survey (SF-36), focusing on domains such as bodily pain, physical functioning, and mental health. Each domain score ranges from 0 to 100, with higher scores indicating better health status. Improvements of ≥5 points in physical functioning or bodily pain subscales will be considered meaningful.

SECONDARY OUTCOMES:
Change in Physical Function | Baseline and Week 12
  Assessed via the 6-Minute Walk Test (6MWT). Participants will be instructed to walk as far as possible on a flat surface for 6 minutes. The total distance (in meters) will be recorded. An increase of ≥30 meters is considered clinically significant in CKD populations.
Rate of changes of balance and fall risk | Baseline and Week 12
  Assessing balance improvements and fall risk reduction using Timed Up and Go (TUG) Test duration (unit: seconds, Time required to rise, walk 3 meters, turn, and return; diagnostic threshold ≥12 seconds indicates fall risk).
Change in Bowel Health | Baseline and Week 12
  Bowel health will be assessed using the Bristol Stool Form Scale (BSFS), a validated 7-point scale that classifies stool consistency and form. Types 3 and 4 are considered ideal, while types 1-2 indicate constipation. Participants will self-report stool type and frequency. Improvement will be defined as a shift toward type 3 or 4 and/or an increase in the frequency of normal bowel movements. The BSFS is commonly used in peritoneal dialysis research to monitor bowel function and identify constipation.

CONTACTS AND LOCATIONS:
Locations (1):
- Pardis specialized wellness institute, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the published article, after deidentification are to be shared
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Not applicable. It will be accessible for public.

REFERENCES:
- [Background] Yi C, Ye H, Lin J, Chang Y, Zhang X, Zhou T, Yang R, Yang X. The incidence of pain and its association with quality of life in patients with peritoneal dialysis. Ren Fail. 2022 Dec;44(1):724-730. doi: 10.1080/0886022X.2022.2068444. PMID 35491880
- [Background] Bdair A, Tamimi R, Shratih A, Abuhalima D, Abdalla M, Sarsour A, Jebreen K, Hamdan Z, Nazzal Z. Assessing pain levels and quality of life in peritoneal dialysis patients: a cross-sectional study. BMC Nephrol. 2025 Mar 27;26(1):155. doi: 10.1186/s12882-025-04083-6. PMID 40148828
- [Background] Aljenaidi H, Alayoobi L, Alqassab W, Alfehaid A, Albuainain M, AlMuhanadi R, Alotaibi S, Almutiri M, Jaradat A, El-Agroudy AE. Quality of Life in Hemodialysis Versus Peritoneal Dialysis Patients in Bahrain. Cureus. 2023 Nov 25;15(11):e49408. doi: 10.7759/cureus.49408. eCollection 2023 Nov. PMID 38149127
- [Background] Jung HY, Jeon Y, Park Y, Kim YS, Kang SW, Yang CW, Kim NH, Choi JY, Cho JH, Park SH, Kim CD, Kim YL. Better Quality of Life of Peritoneal Dialysis compared to Hemodialysis over a Two-year Period after Dialysis Initiation. Sci Rep. 2019 Jul 16;9(1):10266. doi: 10.1038/s41598-019-46744-1. PMID 31312004
- [Background] Sitjar-Suner M, Suner-Soler R, Masia-Plana A, Chirveches-Perez E, Bertran-Noguer C, Fuentes-Pumarola C. Quality of Life and Social Support of People on Peritoneal Dialysis: Mixed Methods Research. Int J Environ Res Public Health. 2020 Jun 14;17(12):4240. doi: 10.3390/ijerph17124240. PMID 32545857
- [Background] Chu EC, Yau K, Yun SMH. Spondylodiscitis in a Patient Undergoing Chronic Peritoneal Dialysis Presenting to a Chiropractor: Case Report and a Review of the Literature. Cureus. 2023 Aug 29;15(8):e44312. doi: 10.7759/cureus.44312. eCollection 2023 Aug. PMID 37779747
- [Background] Kesikburun B, Eksioglu E, Akdag I, Cakci A. Low back pain in hemodialysis patients: Risk factors and its impact on health-related quality of life. Turk J Phys Med Rehabil. 2017 Nov 15;64(1):66-71. doi: 10.5606/tftrd.2018.1016. eCollection 2018 Mar. PMID 31453491
- [Background] Bennett PN, Hussein WF, Matthews K, West M, Smith E, Reiterman M, Alagadan G, Shragge B, Patel J, Schiller BM. An Exercise Program for Peritoneal Dialysis Patients in the United States: A Feasibility Study. Kidney Med. 2020 Mar 17;2(3):267-275. doi: 10.1016/j.xkme.2020.01.005. eCollection 2020 May-Jun. PMID 32734246
- [Background] Mujahid M, Nasir K, Qureshi R, Dhrolia M, Ahmad A. Comparison of the Quality of Sleep in Patients With Chronic Kidney Disease and End-Stage Renal Disease. Cureus. 2022 Apr 5;14(4):e23862. doi: 10.7759/cureus.23862. eCollection 2022 Apr. PMID 35530875
- [Background] Zhang H, Yang Y, Huang J, Lailan S, Tao X. Correlates of objective sleep quality in older peritoneal dialysis patients. Ren Fail. 2021 Dec;43(1):180-187. doi: 10.1080/0886022X.2020.1871369. PMID 33459122
- [Background] Hedayati SS, Minhajuddin AT, Toto RD, Morris DW, Rush AJ. Validation of depression screening scales in patients with CKD. Am J Kidney Dis. 2009 Sep;54(3):433-9. doi: 10.1053/j.ajkd.2009.03.016. Epub 2009 Jun 3. PMID 19493600
- [Background] Halue G, Tharapanich H, Phannajit J, Kanjanabuch T, Banjongjit A, Lorvinitnun P, Sritippayawan S, Sopassathit W, Poonvivatchaikarn U, Buranaosot S, Somboonsilp W, Wongtrakul P, Boonyakrai C, Narenpitak S, Tatiyanupanwong S, Saikong W, Uppamai S, Panyatong S, Chieochanthanakij R, Lounseng N, Wongpiang A, Treamtrakanpon W, Rattanasoonton P, Lukrat N, Songviriyavithaya P, Parinyasiri U, Rojsanga P, Kanjanabuch P, Puapatanakul P, Pongpirul K, Johnson DW, Perl J, Pecoits-Filho R, Ophascharoensuk V, Tungsanga K; Thailand PDOPPS Steering Committee. Constipation and clinical outcomes in peritoneal dialysis: Results from Thailand PDOPPS. Nephrology (Carlton). 2023 Aug;28 Suppl 1:35-47. doi: 10.1111/nep.14224. PMID 37534844